CLINICAL TRIAL: NCT02418650
Title: A Two-Part Open-Label, Single-Centre Mass Balance, Pharmacokinetics, Biotransformation and Absolute Bioavailability Study of ODM-201 in Healthy Male Subjects
Brief Title: Mass Balance, Pharmacokinetics, Biotransformation and Bioavailability Study of ODM-201 in Healthy Male Subjects
Acronym: ARIADME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 3104005
Record Dates: First submitted 2015-03-24; First posted 2015-04-16 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
Keywords: volunteers
MeSH Terms: interventions — darolutamide; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Experimental): A single oral 300 mg tablet of ODM-201 followed by single intravenous 100 microg of 14C-ODM-201 containing not more than 37 kBq (1000 nCi)14C
  Interventions: Drug: ODM-201 300 mg tablet; Drug: intravenous14C-ODM-201
- Part 2 (Experimental): A single oral solution of 300 mg 14C-ODM-201 containing no more than 6.3 MBq (171 microCi) 14C
  Interventions: Drug: 300 mg 14C-ODM-201 oral solution

INTERVENTIONS:
Drug: ODM-201 300 mg tablet
  Arms: Part 1
Drug: intravenous14C-ODM-201
  Arms: Part 1
Drug: 300 mg 14C-ODM-201 oral solution
  Arms: Part 2

SUMMARY:
A study to investigate absolute bioavailability of ODM-201 and to determine the mass balance and routes of excretion of ODM-201 in healthy volunteers.

DETAILED DESCRIPTION:
6 healthy male subjects will be enrolled in part 1 and part 2 of the study, respectively

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy males
* Aged 50 to 65 years (inclusive)
* Normal weight defined as a body mass index (BMI) of >18.5 and <32.0 kg/m2
* Weight 55 to 100 kg (inclusive)
* Adequate method of contraception during the study and for a period of 6 months after study drug administration

Key exclusion Criteria:

* Evidence of clinically significant disease
* Intake of any medication that could affect the outcome of the study
* Known hypersensitivity to the active substances or the excipients of the drug or any serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* History of anaphylactic/anaphylactoid reactions
* Clinically significant abnormal biochemistry, haematology or urinalysis
* Current or history of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
* Current use or use within the last 12 months of nicotine products
* Positive drugs of abuse test result
* Positive hepatitis B surface antigen, hepatitis C virus antibody or human immunodeficiency virus results
* Presence or history of clinically significant allergy requiring treatment

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Amount of 14C-ODM-201 dose excreted and cumulative amount excreted in urine and faeces and total. Amount excreted and cumulative amount excreted in urine, faeces and total expressed as a percentage of the administered dose. | Urine and faecal samples are collected baseline (Day-1) 72 h post-dose after IV dosing and up-to 14 day post-dose after oral solution dosing

OTHER OUTCOMES:
Metabolite profile of 14C-ODM-201 in plasma, urine and faeces | up to 14 days post-dose after oral solution dosing
Maximum concentration (Cmax) of 14C-radioactivity in plasma | The samples were taken 72 h post-dose after IV dosing and up-to 14 day post-dose after oral solution dosing
Time to maximum concentration (tmax) of 14C-radioactivity in plasma | The samples were taken 72 h post-dose after IV dosing and up-to 14 day post-dose after oral solution dosing
Area under the plasma concentration-time curve (AUC(0-t)) of 14C-radioactivity in plasma | The samples were taken 72 h post-dose after IV dosing and up-to 14 day post-dose after oral solution dosing
Area under the plasma concentration-time curve (AUC(0-infinity)) of 14C-radioactivity in plasma | The samples were taken 72 h post-dose after IV dosing and up-to 14 day post-dose after oral solution dosing
Half life (t1/2) of 14C-radioactivity in plasma | The samples were taken 72 h post-dose after IV dosing and up-to 14 day post-dose after oral solution dosing
Maximum concentration (Cmax) of ODM-201 in plasma | The samples were taken 72 h post-dose after IV dosing and up-to 216 h post-dose after oral solution dosing
Time to maximum concentration (tmax) of ODM-201 in plasma | The samples were taken 72 h post-dose after IV dosing and up-to 216 h post-dose after oral solution dosing
Area under the plasma concentration-time curve (AUC(0-t)) of ODM-201 in plasma | The samples were taken 72 h post-dose after IV dosing and up-to 216 h post-dose after oral solution dosing
Area under the plasma concentration-time curve (AUC(0-infinity)) of ODM-201 in plasma | The samples were taken 72 h post-dose after IV dosing and up-to 216 h post-dose after oral solution dosing
Half life (t1/2) of ODM-201 in plasma | The samples were taken 72 h post-dose after IV dosing and up-to 216 h post-dose after oral solution dosing
Maximum concentration (Cmax) of metabolite ORM 15341 in plasma | The samples were taken 72 h post-dose after IV dosing and up-to 216 h post-dose after oral solution dosing
Time to maximum concentration (tmax) of metabolite ORM 15341 in plasma | The samples were taken 72 h post-dose after IV dosing and up-to 216 h post-dose after oral solution dosing
Area under the plasma concentration-time curve (AUC(0-t)) of metabolite ORM 15341 in plasma | The samples were taken 72 h post-dose after IV dosing and up-to 216 h post-dose after oral solution dosing
Area under the plasma concentration-time curve (AUC(0-infinity)) of metabolite ORM 15341 in plasma | The samples were taken 72 h post-dose after IV dosing and up-to 216 h post-dose after oral solution dosing
Half life (t1/2) of metabolite ORM 15341 in plasma | The samples were taken 72 h post-dose after IV dosing and up-to 216 h post-dose after oral solution dosing
Maximum concentration (Cmax) of metabolite 14C-ORM 15341 in plasma | The samples were taken 72 h post-dose after IV dosing
Time to maximum concentration (tmax) of metabolite 14C-ORM 15341 in plasma | The samples were taken 72 h post-dose after IV dosing
Area under the plasma concentration-time curve (AUC(0-t)) of metabolite 14C-ORM 15341 in plasma | The samples were taken 72 h post-dose after IV dosing
Area under the plasma concentration-time curve (AUC(0-infinity)) of metabolite 14C-ORM 15341 in plasma | The samples were taken 72 h post-dose after IV dosing
Half life (t1/2) of metabolite 14C-ORM 15341 in plasma | The samples were taken 72 h post-dose after IV dosing
Maximum concentration (Cmax) of 14C-ODM-201 in plasma | The samples were taken 72 h post-dose after IV dosing
Time to maximum concentration (tmax) of 14C-ODM-201 in plasma | The samples were taken 72 h post-dose after IV dosing
Area under the plasma concentration-time curve (AUC(0-t)) of 14C-ODM-201 in plasma | The samples were taken 72 h post-dose after IV dosing
Area under the plasma concentration-time curve (AUC(0-infinity)) of 14C-ODM-201 in plasma | The samples were taken 72 h post-dose after IV dosing
Half life (t1/2) of 14C-ODM-201 in plasma | The samples were taken 72 h post-dose after IV dosing
Maximum concentration (Cmax) of 14C-radioactivity in whole blood | The samples were taken 24 h post-dose after oral solution dosing
Time to maximum concentration (tmax) of 14C-radioactivity in whole blood | The samples were taken 24 h post-dose after oral solution dosing
Area under the plasma concentration-time curve (AUC(0-t)) of 14C-radioactivity in whole blood | The samples were taken 24 h post-dose after oral solution dosing
Renal elimination for ODM-201 in urine | The samples were taken 72 h post-dose after IV dosing and up-to 14 d post-dose after oral solution dosing
Renal elimination for 14C-ODM-201 in urine | The samples were taken up-to 14 d post-dose after oral solution dosing
Fraction absorbed (FA) of total radioactivity based on urinary recovery of total radioactivity for both IV and oral dosing | The samples were taken 72 h post-dose after IV dosing and up-to 14 d post-dose after oral solution dosing
Adverse events | Collected 7 days post-dose in part 1 and up to 14 days post-dose in part 2
Physical examination | Assessed at screening, pre-dose, at discharge from the study centre (72 h and 7 d post-dose in part 1 and latest at 14 d post-dose in part 2)
  Full physical examination
Blood pressure | Assessed at screening, pre-dose, 3 h, 5 h, 12 h, 24 h, 36 h and 48 h post-dose and at discharge from the study centre (72 h post-dose in part 1 and latest at 14 d post-dose in part 2) and in addition in part 1 7 d post-dose
Heart rate | Assessed at screening, pre-dose, 3 h, 5 h, 12 h, 24 h, 36 h and 48 h post-dose and at discharge from the study centre (72 h post-dose in part 1 and latest at 14 d post-dose in part 2) and in addition in part 1 7 d post-dose
Oral temperature | Assessed at screening, pre-dose, 3 h, 5 h, 12 h, 24 h, 36 h and 48 h post-dose and at discharge from the study centre (72 h post-dose in part 1 and latest at 14 d post-dose in part 2) and in addition in part 1 7 d post-dose
12-lead ECG | Assessed at screening, pre-dose, 3 h, 5 h, 12 h, 24 h, 36 h and 48 h post-dose and at discharge from the study centre (72 h post-dose in part 1 and latest at 14 d post-dose in part 2) and in addition in part 1 7 d post-dose
Clinical chemistry | Assessed at screening, pre-dose, 24 h and 48 h post-dose and 7 d post-dose in part 1 and latest at 14 d post-dose in part 2
  Alanine Aminotransferase, Albumin, Alkaline Phosphatase, Aspartate Aminotransferase, Bilirubin (Total), Calcium, Creatinine, Creatinine clearance, Lactate dehydrogenase, Potassium, Sodium and Urea
Haematology | Assessed at screening, pre-dose, 24 h and 48 h post-dose and 7 d post-dose in part 1 and latest at 14 d post-dose in part 2
  Basophils, Eosinophils, Haematocrit, Haemoglobin, Lymphocytes, MCH, MCHC, MCV, Monocytes, Neutrophils, Red Blood Cell Count, White Blood Cell Count and Thrombocytes
Urinalysis | Assessed at screening, pre-dose, 24 h and 48 h post-dose and 7 d post-dose in part 1 and latest at 14 d post-dose in part 2
  Leucocytes, protein, erythrocytes, glucose and specific gravity

CONTACTS AND LOCATIONS:
Overall Officials: Philip Evans, MB ChB MRCS, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom

REFERENCES:
- [Derived] Zurth C, Nykanen P, Wilkinson G, Taavitsainen P, Vuorela A, Huang F, Reschke S, Koskinen M. Clinical Pharmacokinetics of the Androgen Receptor Inhibitor Darolutamide in Healthy Subjects and Patients with Hepatic or Renal Impairment. Clin Pharmacokinet. 2022 Apr;61(4):565-575. doi: 10.1007/s40262-021-01078-y. Epub 2021 Dec 6. PMID 34866168